CLINICAL TRIAL: NCT00082459
Title: A Randomized Phase II Study Investigating the Route of Administration of Oncophage (HSPPC-96) in Patients With Metastatic Renal Cell Carcinoma
Brief Title: Trial to Compare the Routes of Administration of an Investigational, Personalized, Therapeutic Cancer Vaccine Oncophage (HSPPC-96) in Patients With Metastatic Renal Cell Carcinoma
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Lack of enrollment
Sponsor: Agenus Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: C-100-23
Record Dates: First submitted 2004-05-10; First posted 2004-05-12 (Estimated); Last update posted 2012-09-07 (Estimated); Status verified 2012-09

CONDITIONS: Renal Cell Carcinoma
Keywords: Kidney Cancer; Renal; Tumor; Immunotherapy
MeSH Terms: conditions — Carcinoma, Renal Cell; Kidney Neoplasms; Neoplasms

INTERVENTIONS:
Biological: autologous human tumor-derived HSPPC-96

SUMMARY:
The goal of this trial is to determine the safety of HSPPC-96 and which route of administration achieves a better response with the vaccine. HSPPC-96 is an immunotherapeutic agent made from an individual patient's tumor.

DETAILED DESCRIPTION:
The goal of this trial is to determine the safety of HSPPC-96 and which route of administration achieves a better response with the vaccine. HSPPC-96 is an immunotherapeutic agent made from an individual patient's tumor. The study is being conducted in Houston, Texas with patients enrolled into one of two treatment arms. The two treatment arms are either subcutaneous injection or intradermal injection, both with HSPPC-96. To be treated with HSPPC-96 patients must undergo surgery to remove the kidney tumor and a portion of this tissue will be sent to Antigenics' manufacturing facility for processing.

ELIGIBILITY:
Inclusion Criteria:

* Suspected metastatic renal cell carcinoma (AJCC Stage IV) with intact primary tumor
* No previous therapy for metastatic renal cell carcinoma
* Measurable disease (RECIST criteria)
* Primary tumor greater than or equal to 7cm on CT or MRI
* ECOG performance status 0-1
* At least 18 years old
* Life expectancy > 3 months
* Adequate cardiac function (NYHA I-II)
* Not pregnant
* Provide written informed consent
* Absence of multiple liver metastases, brain or threatening bone metastases (axial skeleton and/or pathological features)
* Planned complete nephrectomy

Exclusion Criteria:

* History of primary or secondary immunodeficiency, or patients using systemic corticosteroids or cyclosporin A
* Other cancer (including renal cell carcinoma) within the last five years (with the exception of adequately treated cone-biopsied in situ carcinoma of the cervix uteri or basal or squamous cell carcinoma of the skin)
* Embolization of the renal artery prior to nephrectomy
* Active, uncontrolled infection or other serious medical illnesses, preventing study completion, in the opinion of the Principal Investigator

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40
Dates: Start 2002-07; Primary Completion 2005-12 (Actual); Study Completion 2005-12 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Houston, Texas, United States